CLINICAL TRIAL: NCT00813046
Title: Preliminary Assessment of the Short Term Clinical Tolerability and Safety of Grass Pollen-derived Peptides for Oral Use in Antigen-specific Immunotherapy of Seasonal Allergic Rhinoconjunctivitis
Brief Title: Safety and Tolerance Study of Grass Pollen-derived Peptides to Treat Allergic Rhinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioTech Tools S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTT-gpASIT002; EudraCT 2008-006368-12
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2014-05-26 (Estimated); Status verified 2014-05

CONDITIONS: Seasonal Allergic Rhinoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gpASIT+TM (Experimental)
  Interventions: Biological: gpASIT+TM

INTERVENTIONS:
Biological: gpASIT+TM — oral administration of entero-coated capsules containing increasing doses of gpASIT+TM (25 to 1600µg), one dose per day for 4 days

SUMMARY:
The purpose of this study is to determine whether the oral administration of grass pollen peptides to treat allergic rhinitis is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years
* The subjects are in good physical and mental health according to his/her medical history, vital signs, and clinical status
* Male or non-pregnant, non-lactating females
* A history of seasonal allergic rhinoconjunctivitis (SAR) during the grass pollen season during at least the last two years
* A positive skin prick test to grass-pollen mixture
* Specific IgE against grass pollen (RAST class 2 or IgE > 0.7 kU/l)
* Asymptomatic to perennial inhalant allergens

Exclusion Criteria:

* Subjects with current or past immunotherapy for SAR
* Subjects requiring controller medication against asthma (bronchodilator nebulised drugs or local or systemic corticosteroids)
* Documented evidence of acute or significant chronic sinusitis (as determined by individual investigator)
* Subjects with a history of food allergy and consecutive anaphylaxis
* Subjects with a history of hepatic or renal disease
* Subject with malignant disease, autoimmune disease
* Female subjects who are pregnant, lactating, or of child-bearing potential and not protected from pregnancy by a sufficiently reliable method (OCs, IUD).
* Females unable to bear children must have documentation of such (i.e. tubal ligation, hysterectomy, or post menopausal [defined as a minimum of one year since the last menstrual period])
* Any chronic disease, which may impair the subject's ability to participate in the trial (i.e. severe congestive heart failure, active gastric or duodenal ulcer, uncontrolled diabetes mellitus, etc…)
* Subjects with clinically relevant abnormal QTc intervals of the ECG : QTc > 450 ms for man and > 470 ms for women
* Subjects requiring beta-blockers medication
* Chronic use of concomitant medications that would affect assessment of the effectiveness of the study medication (e.g. tricyclic antidepressants)
* Subject with febrile illness (> 37.5°C, oral)
* A known positive serology for HIV-1/2, HBs antigen or anti-HCV antibodies
* The subject is immunocompromised by medication or illness, has received a vaccine, corticoids or immunosuppressive medications within 1 month before study entry
* Receipt of blood or a blood derivative in the past 6 months preceding study entry
* Regular consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 4 weeks preceding the study, any consumption of corticoids (oral, topic or nasal) or of anti-histaminic drugs within 1 week preceding the study
* Use of long-acting antihistamines
* Any condition which could be incompatible with protocol understanding and compliance
* Subjects who have forfeited their freedom by administrative or legal award or who are under guardianship,
* Participation in another clinical trial and/or treatment with an experimental drug within 1 month of study start
* A history of hypersensitivity to the excipients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To demonstrate the clinical tolerability and safety of the treatment by looking at the absence of immediate allergic reaction. | 10 days

SECONDARY OUTCOMES:
vital signs clinical laboratory evaluations adverse events general physical status | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital University Ghent, Ghent, Belgium